CLINICAL TRIAL: NCT05694572
Title: Post-market Surveillance of Micorport CRM Cardiac Implantable Electronic Devices
Acronym: PIANO
Status: Recruiting | Type: Observational
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: LMIO01
Record Dates: First submitted 2022-12-20; First posted 2023-01-23 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Rhythm Disorder; Heart Failure; Sudden Cardiac Death
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pacemaker system: Patients implanted with ENO or ALIZEA family pacing systems
  Interventions: Device: Implantation of a CIED
- ICD system: Patients implanted with ULYS family ICD systems
  Interventions: Device: Implantation of a CIED
- CRT-D system: Patients implanted with GALI family CRT-D systems
  Interventions: Device: Implantation of a CIED

INTERVENTIONS:
Device: Implantation of a CIED — Implantation of a CIED

SUMMARY:
The primary objective of the study is to assess the chronic safety of MicroPort CRM market-released systems.

DETAILED DESCRIPTION:
PIANO Post Market Surveillance (PMS) investigation will cover MicroPort CRM systems CE- market and released since 2018.

Continuous monitoring of MicroPort CRM market-released systems will also enable to:

* confirm the safety and performance of the device throughout the study duration
* identify previously unknown side-effects and monitoring the identified side-effects and contraindications,
* identify and analyse emergent risks on the basis of factual evidence, ensuring the continued acceptability of the benefit-risk ratio
* identify possible systematic misuse or off-label use of the device, with a view to verifying that the intended purpose is correct

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria at the time of the inclusion visit may be enrolled in the study:

1. Subject implanted with one of the following MicroPort CRM market-released system:

   * ENO, TEO, OTO, ALIZEA, BOREA, or CELEA PM single chamber (SR) or dual chamber (DR) implanted after 01 January 2020 in combination with at least one XFINE or VEGA pacing lead
   * ULYS, EDIS ICD single chamber (VR) or dual chamber (DR) system in combination with an INVICTA defibrillation lead. Additional XFINE or VEGA atrial pacing lead is optional.
   * GALI CRT-D implanted in combination with an INVICTA defibrillation lead. Additional NAVIGO left ventricular pacing lead is optional.
   * GALI SONR CRT-D in combination with an INVICTA defibrillation lead and with either a NAVIGO left ventricular or a SONRTIP atrial pacing lead.
   * Future generation of market approved MicroPort CRM PM, ICD or CRT-D device associated with existing or future generation of MicroPort CRM lead
2. Subject equipped with Remote Monitoring System (RMS) (only for subject implanted with ICD or CRT-D system)
3. Subject followed yearly per standard practice by investigational site: in-clinic visit or remote visit through remote monitoring system
4. Subject reviewed, signed and dated the Informed Consent Form (ICF) if applicable per country regulation

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to be enrolled in the study:

1. Age less than 18 years old or more than 90 years at time of inclusion, incapacitated or under guardianship or kept in detention
2. Life expectancy less than 1 year
3. Currently enrolled in an active study of MicroPort CRM

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects implanted with a pacemaker, an Implantable Cardioverter-Defibrillator (ICD) or a Cardiac Resynchronization Therapy (CRT-D) Class I or II indication according to the latest guidelines from the European Society of Cardiology (ESC)1 or from the American College of Cardiology (ACC)/ American Heart Association (AHA)/ Heart Rhythm society (HRS)2 as appropriate per geography.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2031-06-15 (Estimated); Study Completion 2031-06-15 (Estimated)

PRIMARY OUTCOMES:
Chronic complication free rate of MicroPort CRM market-released system | Through study duration, an average of 5 years
  Complications are defined as device-related reinterventions or deaths

SECONDARY OUTCOMES:
Acute complication free rate | Up to 3 months post-implant
  Complications are defined as device-related reinterventions or deaths
Overall complication free rate | Through study duration, an average of 5 years
  Complications are defined as device-related reinterventions or deaths
Annual complication free rate | Through study duration, an average of 1 year
  Complications are defined as device-related reinterventions or deaths

CONTACTS AND LOCATIONS:
Overall Officials: Yann POEZEVARA, MSc, Study Director — MicroPort CRM
Locations (1):
- Hospital Santa Marta Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided